CLINICAL TRIAL: NCT00791596
Title: Effectiveness of an Ergonomic Intervention on Work-Related Posture and Low Back Pain in Video Display Terminal Operators: a 3 Year Cross-Over Trial
Brief Title: Effectiveness of Ergonomic Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Paolo Pillastrini, University of Bologna
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PP001012008
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-10

CONDITIONS: Low Back Pain; Neck Pain; Upper Extremity; Lower Extremity
Keywords: Ergonomic intervention; Musculoskeletal disorders; Low back pain; Posture; Video display terminal
MeSH Terms: conditions — Low Back Pain; Neck Pain; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): The first Arm received the intervention between baseline and the first follow-up, whereas the second Arm was the Control group
  Interventions: Other: Ergonomic Intervention
- 2 (Experimental): The second Arm received the intervention between the third and the fourth follow-up, whereas the first Arm was the Control group
  Interventions: Other: Ergonomic Intervention

INTERVENTIONS:
Other: Ergonomic Intervention — The intervention used in this investigation was an ergonomic adjustment of the VDT workstation design
  Other Names: Preventive Intervention of Musculoskeletal Disorders

SUMMARY:
This Research study aims to investigate the long term effectiveness of a workstation ergonomic intervention for work-related posture and low back pain (LBP) of Video Display Terminal (VDT) workers

DETAILED DESCRIPTION:
A non-randomized, crossover trial design was used with follow-up repeated 6, 12, and 30 months from baseline in the first intervention period and then beginning at 6 months following the crossover.

The administrative offices in the two main buildings of the town hall of Forlì, Italy.

The study population was composed of 400 employees, who used VDTs for at least 20 hours a week, of whom we randomly selected 100 participants from each building. Of the 200 initial participants, 153 completed the study; the dropouts were due to illness/injury or maternity.

Participants were assigned to intervention or control during the first period and then crossed over after a 30-month washout. The intervention used in this investigation was an ergonomic adjustment of the VDT workstation design.

Our study showed that the workstation ergonomic adjustment improved work-related posture and in reducing LBP in VDT operators among subjects who received the intervention both in the first period and in the crossover, and maintained these positive effects for at least 30 months.

ELIGIBILITY:
Inclusion Criteria:

* The study population was composed of 400 employees, who used VDTs for at least 20 hours a week

Exclusion Criteria:

* Subjects were excluded if pregnant or had a medical history of serious injury, spinal surgery, malignant pathology, or severe disability

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-01; Primary Completion 2005-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
R.E.B.A. (Rapid Entire Body Assessment) method | Baseline, 6 months, 12 months, 30 months, 36 months

SECONDARY OUTCOMES:
Pain Drawing with a Visual Analogue Scale | Baseline, 6 months, 12 months, 30 months, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pillastrini, MSc, Principal Investigator — University of Bologna
Locations (1):
- University of Bologna, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Result] Pillastrini P, Mugnai R, Farneti C, Bertozzi L, Bonfiglioli R, Curti S, Mattioli S, Violante FS. Evaluation of two preventive interventions for reducing musculoskeletal complaints in operators of video display terminals. Phys Ther. 2007 May;87(5):536-44. doi: 10.2522/ptj.20060092. Epub 2007 Apr 3. PMID 17405805
- [Derived] Pillastrini P, Mugnai R, Bertozzi L, Costi S, Curti S, Guccione A, Mattioli S, Violante FS. Effectiveness of an ergonomic intervention on work-related posture and low back pain in video display terminal operators: a 3 year cross-over trial. Appl Ergon. 2010 May;41(3):436-43. doi: 10.1016/j.apergo.2009.09.008. Epub 2009 Oct 23. PMID 19853837